CLINICAL TRIAL: NCT02711202
Title: A Pilot, Open Single Centre, Prospective, Parallel Trail to Evaluate the Efficacy and Safety of Immunosuppressive Regimen Without Calcineurin Inhibitors and Steroids After Induction of Anti-CD52 and Anti-TNF-α Monoclonal Antibodies in Kidney Transplant Recipients
Brief Title: Sequential Targeting of Cluster of Differentiation 52 (CD52) and Tumor Necrosis Factor (TNF) Allows Early Minimization Therapy in Kidney Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Collaborators: Charite University, Berlin, Germany (Other); Miltenyi Biomedicine GmbH (Industry)
Responsible Party: Principal Investigator, Petra Hruba, IKEM, Institute for Clinical and Experimental Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: EudraCT Number: 2006-003110-18
Record Dates: First submitted 2016-03-09; First posted 2016-03-17 (Estimated); Results first posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Alemtuzumab; Infliximab; Sirolimus; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sirolimus (Active Comparator): Patients received two applications of anti-CD52 MabCampath (Alemtuzumab), a single dose of anti-TNF-α Remicade (Infliximab) monoclonal antibodies in the early posttransplant period. First 14 days patients received tacrolimus monotherapy, at post-operative day (POD) 14, they were randomized to sirolimus monotherapy.
  Interventions: Drug: MabCampath,; Drug: Remicade; Drug: Sirolimus; Drug: Tacrolimus
- Tacrolimus (Active Comparator): Patients received two applications of anti-CD52 MabCampath (Alemtuzumab), a single dose of anti-TNF-α Remicade (Infliximab) monoclonal antibodies in the early posttransplant period. First 14 days patients received tacrolimus monotherapy, at POD 14, they were randomized to tacrolimus monotherapy.
  Interventions: Drug: MabCampath,; Drug: Remicade; Drug: Tacrolimus

INTERVENTIONS:
Drug: MabCampath, — Primary deceased donor kidney transplant recipients received 2x20 mg Alemtuzumab (day 0/day 1) followed by 5 mg/kg Infliximab (day 2). For 14 days all patients received only tacrolimus, then they were randomized to either receive tacrolimus (TAC, n=13) or sirolimus (SIR, n=7) monotherapy, respectively.
  Other Names: Alemtuzumab
Drug: Remicade — Primary deceased donor kidney transplant recipients received 2x20 mg Alemtuzumab (day 0/day 1) followed by 5 mg/kg Infliximab (day2). For 14 days all patients received only tacrolimus, then they were randomized to either receive tacrolimus (TAC, n=13) or sirolimus (SIR, n=7) monotherapy, respectively.
  Other Names: Infliximab
Drug: Sirolimus — Primary deceased donor kidney transplant recipients received 2x20 mg Alemtuzumab (day 0/day 1) followed by 5 mg/kg Infliximab (day 2). For 14 days all patients received only tacrolimus, then they were randomized to either receive tacrolimus (TAC, n=13) or sirolimus (SIR, n=7) monotherapy, respectively.
  Arms: Sirolimus
Drug: Tacrolimus — Primary deceased donor kidney transplant recipients received 2x20 mg Alemtuzumab (day 0/day 1) followed by 5 mg/kg Infliximab (day 2). For 14 days all patients received only tacrolimus, then they were randomized to either receive tacrolimus (TAC, n=13) or sirolimus (SIR, n=7) monotherapy, respectively.

SUMMARY:
The aim of the study is to evaluate the efficacy of new immunosuppressive protocol based on two applications of anti-CD52 MabCampath (Alemtuzumab) a single dose of anti-TNF-α Remicade (infliximab) monoclonal antibodies in the early posttransplant period followed by either monotherapy based on tacrolimus or sirolimus.

ELIGIBILITY:
Inclusion criteria:

* First deceased-donor kidney transplantation
* Age >18 years
* Donor <65 years
* Cytomegalovirus (CMV)/ Epstein-Barr virus (EBV) seropositivity
* panel reactive antibodies (PRA) <10%
* Written consent

Exclusion criteria:

* Retransplantation, combined transplantation
* Prior immunosuppression less than 6 months prior transplantation
* Induction therapy with antibodies
* Leukopenia < 4000, thrombocytopenia < 100 000, Haemoglobin < 80 g/l
* History of antithymoglobulin (ATG) or anti-cluster of differentiation 3 (CD3) monoclonals or anti-TNF-α
* Tuberculosis history
* Anti-hepatitis C virus (HCV) positivity, HBsAg
* HIV positivity
* Malignancy history
* Allergy to study medication
* Fertile women without contraception
* Pregnancy, breastfeeding mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ondrej Viklicky, M.D.,Prof., Principal Investigator — Institute for Clinical and Experimental Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Viklicky O, Hruba P, Tomiuk S, Schmitz S, Gerstmayer B, Sawitzki B, Miqueu P, Mrazova P, Tycova I, Svobodova E, Honsova E, Janssen U, Volk HD, Reinke P. Sequential Targeting of CD52 and TNF Allows Early Minimization Therapy in Kidney Transplantation: From a Biomarker to Targeting in a Proof-Of-Concept Trial. PLoS One. 2017 Jan 13;12(1):e0169624. doi: 10.1371/journal.pone.0169624. eCollection 2017. PMID 28085915
- See also: Sequential Targeting of CD52 and TNF Allows Early Minimization Therapy in Kidney Transplantation: From a Biomarker to Targeting in a Proof-Of-Concept Trial — https://pubmed.ncbi.nlm.nih.gov/28085915/
- See also: GEO accession for microarray data for peripheral blodd gene expression — http://www.ncbi.nlm.nih.gov/geo/query/acc.cgi?token=rrctnosmwwkoavs&acc=GSE39299).

RESULTS

PARTICIPANT FLOW:
Groups:
- Sirolimus: Patients received two applications of anti-CD52 MabCampath (Alemtuzumab), a single dose of anti-TNF-α Remicade (Infliximab) monoclonal antibodies in the early posttransplant period. First 14 days patients received tacrolimus monotherapy, at post-operative day (POD) 14, they were randomized to sirolimus monotherapy.
  MabCampath,: Primary deceased donor kidney transplant recipients received 2x20 mg Alemtuzumab (day 0/day 1) followed by 5 mg/kg Infliximab (day 2). For 14 days all patients received only tacrolimus, then they were randomized to sirolimus monotherapy.
- Tacrolimus: Patients received two applications of anti-CD52 MabCampath (Alemtuzumab), a single dose of anti-TNF-α Remicade (Infliximab) monoclonal antibodies in the early posttransplant period. First 14 days patients received tacrolimus monotherapy, at POD 14, they were randomized to tacrolimus monotherapy.
  MabCampath: Primary deceased donor kidney transplant recipients received 2x20 mg Alemtuzumab (day 0/day 1) followed by 5 mg/kg Infliximab (day 2). For 14 days all patients received only tacrolimus, then they were randomized to tacrolimus monotherapy.
Period: Overall Study
Arm/Group | Sirolimus | Tacrolimus
Started | 7 | 13
Completed | 3 | 13
Not Completed | 4 | 0
Not completed — Adverse Event | 3 | 0
Not completed — graft loss | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sirolimus | Tacrolimus | Total
Number analyzed (Participants) | 7 | 13 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 12 | 19
  >=65 years | 0 | 1 | 1
Age, Continuous [Median (Full Range); unit: years] | 46 [29 to 55] | 55 [20 to 70] | 51 [20 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 5 | 8 | 13
Region of Enrollment [Number; unit: participants]
  Czechia | 7 | 13 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Alive
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 7 | 13
Participants | 7 | 13

2. Primary Outcome: Number of Patients With Functional Graft
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 7 | 13
Participants | 6 | 13

3. Secondary Outcome: Kidney Graft Function (Measured by Serum Creatinine)
Description: Kidney graft function is measured as serum creatinine in umol/l at 1 year after transplantation. Higher levels of creatinine represents worse graft function.
Time Frame: 1 year
Measure: Median (Full Range); unit: µmol/l
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 7 | 13
µmol/l | 144.4 [86 to 271.1] | 110 [79.8 to 200.2]

4. Secondary Outcome: Number of Bioptically Verified Rejection Episodes
Description: We calculated the number of participants with biopsy-proven subclinical rejection (based on Banff classification) within 1 year post-transplantation.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 7 | 13
Participants | 4 | 2

5. Secondary Outcome: Presence of Subclinical Rejection in Protocol Biopsy at 12 Months (Based on Histological Examination Using Banff Classification)
Time Frame: 1 year
Population: In Sirolimus arm, 12 months protocol biopsy has not been performed in 2 patients
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 7 | 13
Participants | 1 | 2

ADVERSE EVENTS:
Arm/Group | Sirolimus | Tacrolimus
Serious Adverse Events (participants affected / at risk) | 5/7 | 0/13
Other Adverse Events (participants affected / at risk) | 5/7 | 9/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sirolimus (N=7) | Tacrolimus (N=13)
Proteinuria (Renal and urinary disorders) | 5 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus (N=7) | Tacrolimus (N=13)
Infections (Infections and infestations) | 5 (5) | 9 (9)
cardio vascular disorders (Cardiac disorders) | 2 (2) | 3 (3) — ischemic cardiac desease stroke
Delayed graft function (Renal and urinary disorders) | 1 (1) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Hyperparathyreosis (Metabolism and nutrition disorders) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes